CLINICAL TRIAL: NCT03856099
Title: A Multicenter, Open-Label, Phase Ⅱ Clinical Trial to Evaluate the Safety and Efficacy of TTAC-0001, a Fully Human Monoclonal Antibody in Patients With Recurrent Glioblastoma Progressed on Bevacizumab Including Therapy
Brief Title: TTAC-0001 Phase II Trial With Recurrent Glioblastoma Progressed on Bevacizumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Subject recruitment issues and follow-up study plans
Sponsor: PharmAbcine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PMC_TTAC-0001_03
Record Dates: First submitted 2019-02-21; First posted 2019-02-27 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — olinvacimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TTAC-0001 (Experimental): TTAC-0001 with dose assigned to each dose group will be administered
  Interventions: Drug: TTAC-0001

INTERVENTIONS:
Drug: TTAC-0001 — * Investigational product (IP): TTAC-0001
  * Treatment groups: 3 dose groups
    * Dose group A : TTAC-0001 16 mg/kg on D1 and D15
    * Dose group B : TTAC-0001 20 mg/kg on D1 and D15
    * Dose group C : TTAC-0001 24 mg/kg on D1 and D15
  * Cycle: 4 weeks (28 days per cycle)

SUMMARY:
This is a phase II, open-Label clinical trial to evaluate the safety and efficacy of TTAC-0001 in patients with recurrent glioblastoma who was progressed on bevacizumab including therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent prior to any study specific procedures, sampling or analyses.
2. Aged at least 18 years old
3. Patients must have a histologically proven diagnosis of glioblastoma/gliosarcoma
4. Patients must have previous treatment including bevacizumab
5. Patients must have a radiological diagnosis of recurrent/relapsed or progressive glioblastoma/gliosarcoma after bevacizumab including therapy according to response assessment in neuro-oncology (RANO) criteria
6. At least one confirmed measurable lesion or non measurable lesion as determined by RANO criteria
7. Patients must undergo IDH1 mutational testing on a tumor specimen before entering the study. Immunohistochemistry (IHC) is sufficient for enrollment, although DNA sequencing may also be performed as per local institutional guidelines. Patients are eligible regardless of their tumor status.
8. Karnofsky Performance Status (KPS) ≥ 70
9. A person who satisfies the following criteria in hematologic, renal, and hepatic function tests (1) Hematologic tests - Absolute neutrophil count (ANC) ≥ 1.5 x 109/L - Platelets ≥ 75 x 109/L

   - Hemoglobin ≥ 9.0 g/dL (2) Blood coagulation tests

   - Prothrombin time (PT) ≤ 1.5 x Upper limit of normal (ULN)

   - Activated partial thromboplastin Time (aPTT) ≤ 1.5 x ULN (3) Hepatic function tests
   * Total bilirubin ≤ 1.5 x ULN
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 x ULN (4) Renal function test
   * Creatinine clearance (CrCl) ≥ 30 mL/minute calculated by Cockcroft-Gault formula
10. Life expectancy of at least 12 weeks
11. Females of child bearing potential must have a negative pregnancy test during screening and must not be breastfeeding or intending to become pregnant during the study.
12. Male patients with female partners of child-bearing potential must be willing to use two forms of acceptable contraception, including one barrier method, during their participation in this study and for 16 weeks following the last dose of the study. Refer to section 10.5.1 Restrictions, permitted methods of contraception and definitions.

Exclusion Criteria:

1. Diagnosed with malignant tumors, except basal cell carcinoma, cutaneous squamous cell carcinoma, and noninvasive uterine cervical cancer treated within 2 years prior to receiving the first dose of treatment.
2. The following concomitant diseases:

(1) Uncontrolled hypertension (systolic blood pressure [SBP] > 150 or diastolic blood pressure [DBP] > 90 mmHg) (2) Uncontrolled seizures (3) Class III or IV heart failure according to New York Heart Association (NYHA) classification (4) Oxygen-dependent chronic disease (5) Active psychiatric disorder (schizophrenia, major depressive disorder, bipolar disorder etc.). Treated depression with ongoing antidepressant medication is not an exclusion.

3) Not recovered from AEs < National Cancer Institute -Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade 2 caused by CCRT 4) Treatment with bevacizumab including therapy 2 weeks prior to receiving the first dose of treatment.

5) Undergone major surgery requiring general anesthesia or a respiratory assistance device within 4 weeks prior to the baseline visit (within 2 weeks for video-assisted thoracoscopic surgery [VATS] or open-and-closed [ONC] surgery) 6) Treated with other investigational products within 4 weeks prior to the patient receiving the first dose of treatment.

7) A known history of severe drug hypersensitivity or hypersensitivity to a therapy similar to the study drug 8) Unable to participate in the trial according to the investigator's decision. 9) Patient not eligible for sequential MRI evaluations are not eligible for this study 10) Previous therapy with VEGF-targeted agents except bevacizumab. 11) Known active hepatitis B or hepatitis C infection 12) Has received a live vaccine within 30 days prior to enrollment. Seasonal flu vaccines that do not contain live virus are permitted.

13) Has had a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events | until time of progressive disease or 1 year
  The frequency and percentage of AEs will be presented by dose goup

SECONDARY OUTCOMES:
Progression free survival rate at 4 months | at the end of 4 months
  The rate and 2-sided 95% confidence interval of progression free survival at the 4-month
Progression free survival rate at 6 months | at the end of 6 months
  The rate and 2-sided 95% confidence interval of progression free survival at the 6-month
Progression free survival | until time of progressive disease or time point of patients' death which come first assessed up to 1 year
  Period from the date of the drug administration to the disease progression time point
Overall survival | until time point of patients' death up to 1 year
  Period from the date of the drug administration to the time point of patient's death
Objective response rate | At every 2nd cycles until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year (every cycle is 28 days)
  complete response (CR) or partial response (PR) by RANO criteria
Disease control rate | At every 2nd cycles until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year (every cycle is 28 days)
  complete response (CR), partial response (PR) or stable disease (SD) by RANO criteria

OTHER OUTCOMES:
Immunogenicity | From screening visit to end of treatment visit (time of progressive disease or 1 year)
  Presence anti-drug antibody (ADA)
Pharmacokinetic parameters - Cmax | From screening visit to end of treatment visit (time of progressive disease or 1 year)
  Maximum concentration of drug by dose level
Pharmacokinetic parameters - Cmin | From screening visit to end of treatment visit (time of progressive disease or 1 year)
  Minimum concentration of drug by dose level
Pharmacokinetic parameters - AUC0-t | From screening visit to end of treatment visit (time of progressive disease or 1 year)
  Area under the curve from baseline to each timepoint by dose level
Pharmacokinetic parameters -Tmax | From screening visit to end of treatment visit (time of progressive disease or 1 year)
  Time of Cmax by dose level
Pharmacokinetic parameters - CL | From screening visit to end of treatment visit (time of progressive disease or 1 year)
  Clearance by dose level
Pharmacokinetic parameters - Vd | From screening visit to end of treatment visit (time of progressive disease or 1 year)
  Volume of distribution by dose level
Pharmacokinetic parameters - Ke | From screening visit to end of treatment visit (time of progressive disease or 1 year)
  Elimination rate constant by dose level
Pharmacokinetic parameters - T½ | From screening visit to end of treatment visit (time of progressive disease or 1 year)
  Half-life by dose level
Change in concentration of serum angiogenic factor or receptor | From screening visit to end of treatment visit (time of progressive disease or 1 year)
  VEGF, placental growth factor [PLGF], soluble vascular endothelial growth factor receptor [sVEGFR]-2, sVEGFR-1, etc.
DCE-MRI | Screening visit, on Day8 and Day 15 of cycle 1, Day 28 of every 2nd cycle (1 cycle is 28 days, up to 1 year)
  Blood flow parameter - iAUC, K-trans

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Stanford Avanced Medical Center, Stanford, California
  - Florida Hospital Cancer Institute & Florida Hospital Orlando, Orlando, Florida
- Austin Hospital, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No